CLINICAL TRIAL: NCT05028699
Title: Effect of Common Bean Baked Snack (Phaseolus Vulgaris L.) Consumption on Blood Lipid Levels and Hormones Regulating Appetite and Satiety: Randomized Crossover Clinical Trials
Brief Title: Evaluation of Common Bean Baked Snack Consumption on Blood Lipids in Overweight People With Altered Blood Lipid Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: Centro de Investigación y Asistencia en Tecnología y Diseño del Estado de Jalisco (Unknown)
Responsible Party: Principal Investigator, Alejandro Escobedo Avila, Principal Investigator, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CI-09620
Record Dates: First submitted 2021-08-20; First posted 2021-08-31 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Dyslipidemias
Keywords: Functional food; Common bean; Snack
MeSH Terms: conditions — Dyslipidemias | interventions — Snacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snack (Experimental): 32 g of a common bean baked snack per day for 28 days.
  Interventions: Other: Snack
- Control (No Intervention)

INTERVENTIONS:
Other: Snack — Participants will consume 32 g of a common bean baked snack per day for 28 days during the intervention stage.
  Arms: Snack

SUMMARY:
Introduction: The Mexican population consumes vegetables and snacks with the same frequency. Besides, most of the snacks available on the market contain high fat, sodium and calorie, and low protein levels. Regular consumption of these snacks and low physical activity could promote the development of noncommunicable diseases. Common bean-based snacks are potential healthier alternatives to replace conventional snacks.

Hypothesis: The consumption of a common bean baked snack (Phaseolus vulgaris L.) reduces blood lipid levels in overweight people with altered blood lipid levels.

Objectives: Evaluate the effect of common bean baked snack consumption on blood lipid levels in overweight people with altered blood lipid levels.

Material and Methods: Randomized crossover clinical trial, 28 patients with altered blood lipid levels, 18-40 years old, snack supplementation for four weeks, clinical and laboratory determinations, such as total cholesterol, triglycerides, LDL, HDL, among others.

* Intervention phase: Common bean baked snack intervention.
* Control phase B: No intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25.0 and 29.9 kg/m2,
* Abnormal serum lipid levels:

  * Total cholesterol: ≥200 mg/dL,
  * Low-density lipoproteins: 100 to 190 mg/dL,
  * High-density lipoproteins: <50 mg/dL in females and <40 mg/dL in males,
  * Triglycerides: 150 to 500 mg/dL.

Exclusion Criteria:

* Pregnancy or lactation,
* Plans to lose or gain weight in the next three months,
* Modification of diet or physical activity in the last three months,
* Diagnosis of diabetes, cancer, hypertension, heart disease, gastrointestinal disorder, pancreatitis, kidney, liver or thyroid disease,
* Smoking or drug use,
* Sensitivity for bean consumption,
* Pharmacological treatment or consumption of non-prescription drugs, herbal or nutritional supplements known to modify serum lipid levels.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean low-density lipoprotein (mg/dL) at 28 days | Baseline and 28 days
Change from baseline in the mean high-density lipoprotein (mg/dL) at 28 days | Baseline and 28 days
Change from baseline in the mean total cholesterol (mg/dL) at 28 days | Baseline and 28 days
Change from baseline in the mean triglycerides (mg/dL) at 28 days | Baseline and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Edgar A. Rivera León, PhD, Principal Investigator — Departamento de Biología Molecular y Genómica, Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara
Locations (1):
- Departamento de Biología Molecular y Genómica, Centro Universitario de Ciencias de la Salud, Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
Non-shareable data.